CLINICAL TRIAL: NCT01385735
Title: Effects of Azilect (Rasagiline) on Processing of Emotions, Mood and Executive Function in Parkinson's Disease
Brief Title: Emotion, Mood and Executive Function in Parkinson's Disease (PD)
Acronym: RasQ
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Josef Hospital Bochum (Other)
Responsible Party: Woitalla, Dirk MD, Neurologische Universitätsklinik der Ruhr-Universität Bochum
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2011-TevAzi
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Emotion; mood; executive function
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo 1 Tbl per day, 12 week (84 days) duration
  Interventions: Drug: Placebo
- Rasagiline (Active Comparator): Azilect Group: Dose: 1 mg per day, 12 week (84 days) duration
  Interventions: Drug: Rasagiline

INTERVENTIONS:
Drug: Rasagiline — Azilect Group: Dose: 1 mg per day, 12 week (84 days) duration
  Other Names: Azilect EU/1/04/304/001-007
  Arms: Rasagiline
Drug: Placebo — Placebo 1 Tbl per day, 12 week (84 days) duration
  Arms: Placebo

SUMMARY:
The current study aims to assess the effect of an 8 week Azilect treatment (as adjunct therapy to levodopa) on affect perception and emotional expressiveness in a double-blind placebo-controlled study.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is associated with a range of cognitive impairments, most notably deficits of higher order cognitive control mechanisms referred to as "executive dysfunction". These problems have consistently been related to dysfunction of fronto-striatal circuitry (summary see Stocchi & Brusa, 2000). Executive function impairments may already be present in early stages of PD (Uekermann et al., 2004) and their severity may be exacerbated by affective changes such as depression (Uekermann et al., 2003). In addition to cognitive problems, PD patients frequently suffer from mood changes, in particular apathy (Kirsch-Darrow et al., 2006) and from affect processing impairments, relating to both the ability to decode the affective state of other people on the basis of facial expressions or prosody and to the ability to adequately express the patients' own emotions (e.g. Breitenstein et al., 1998; Zgaljardic et al., 2003, Pell & Leonard, 2005). The capacity for emotion perception was found to be linked to the severity of executive dysfunction; affective and cognitive changes are thus not independent, at least in patients with moderate PD (Breitenstein et al., 2001).

In a recent drug monitoring study by Lundbeck GmbH/TEVA Pharma GmbH based on a small group of PD patients (n=29), introduction of Azilect (Rasagiline) therapy was associated with a significant improvement of PD patients' emotional expressiveness (e.g. facial expression, gestures, voice intonation) over an 8 week observation period. Significant improvements were observed for self-ratings of emotional expressiveness as well as ratings by physicians and relatives. The lack of a placebo-control group, however, does not allow any firm conclusions with regard to the specificity of these effects.

Intact affect recognition and an adequate ability to express emotions are of critical importance for social interaction. The therapeutic efficacy of drug treatment on non-motor symptoms in PD has so far only rarely been addressed. The documentation of a beneficial effect of Azilect on emotional processing would be of great relevance for the quality of life of PD patients and greatly enhance their ability to participate in social life.

The addition of a placebo control group is critical for the assessment of the specificity of the expected beneficial effects of Azilect.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic PD
* age range 30-75 yrs, HY I-III
* stable medication for at least 4 weeks prior to baseline
* Native speakers (German)
* signing of informed consent form

Exclusion Criteria:

* clinically significant depression (BDI>13)
* freezing, pronounced fluctuations
* other neurological or psychiatric disorders
* dementia (MMSE<25)
* treatment with the MAO-B-inhibitor Selegiline, antidepressants
* any contraindication according to SmPC
* participation in another interventional study

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-10 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of Azilect on mood, recognition of facial and vocal affect and emotional expressiveness | 12 weeks
  * Discrimination Faces
  * Discrimination Affect
  * Affect Naming -Faces
  * Discrimination linguistic prosody
  * Discrimination affective prosody
  * Affect naming -congruent and incongruent affective prosody Visual Analogue Scales of emotional expressiveness
  * Rating by study physician and relative
  * Self-rating by patient Assessment of executive function
  * Working Memory (n-back task, digit backward)
  * Verbal Fluency (Regensburger Wortflüssigkeitstest) Beck Depression Inventary (BDI) Apathie Evaluations-Skala (AES) Social Activity Scale - self assessment PDQ-39- self-assessment

SECONDARY OUTCOMES:
Effect on motor function in PD | 12 weeks
  Unified Parkinson's Disease Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- St. Josef Hospital, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Roca M, Torralva T, Gleichgerrcht E, Chade A, Arevalo GG, Gershanik O, Manes F. Impairments in social cognition in early medicated and unmedicated Parkinson disease. Cogn Behav Neurol. 2010 Sep;23(3):152-8. doi: 10.1097/WNN.0b013e3181e078de. PMID 20829664
- [Background] Rosenthal E, Brennan L, Xie S, Hurtig H, Milber J, Weintraub D, Karlawish J, Siderowf A. Association between cognition and function in patients with Parkinson disease with and without dementia. Mov Disord. 2010 Jul 15;25(9):1170-6. doi: 10.1002/mds.23073. PMID 20310053
- [Background] Scholtissen B, Verhey FR, Adam JJ, Weber W, Leentjens AF. Challenging the serotonergic system in Parkinson disease patients: effects on cognition, mood, and motor performance. Clin Neuropharmacol. 2006 Sep-Oct;29(5):276-85. doi: 10.1097/01.WNF.0000229013.95927.C7. PMID 16960473
- [Background] Growdon JH, Kieburtz K, McDermott MP, Panisset M, Friedman JH. Levodopa improves motor function without impairing cognition in mild non-demented Parkinson's disease patients. Parkinson Study Group. Neurology. 1998 May;50(5):1327-31. doi: 10.1212/wnl.50.5.1327. PMID 9595982
- [Background] Timmann D, Daum I. How consistent are cognitive impairments in patients with cerebellar disorders? Behav Neurol. 2010;23(1-2):81-100. doi: 10.3233/BEN-2010-0271. PMID 20714063